CLINICAL TRIAL: NCT01787721
Title: Effect of Manipulation of the Tibiotalar Joint on Gait
Brief Title: Effect of Manipulation of the Ankle Joint on Gait
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit more than 2 subjects
Sponsor: University of Bridgeport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UB-SMP-001
Record Dates: First submitted 2012-11-05; First posted 2013-02-11 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Gait
Keywords: Gait; Ankle joint; Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ankle manipulation (Experimental): Treatment will consist of manipulation of the tibiotalar joint intended to produce anterior to posterior glide of the tibia on the talus
  Interventions: Procedure: Ankle manipulation
- Sham manipulation (Sham Comparator): Sham manipulative procedure of the tibiotalar joint.
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Procedure: Ankle manipulation
  Arms: Ankle manipulation
Other: Sham manipulation
  Arms: Sham manipulation

SUMMARY:
The purpose of this study is to determine if manipulation of the ankle improves some measurable characteristics of how a person walks. The investigators hypothesize that the ankle will be able to bend better after manipulation and thus improve walking speed and reduce differences between the two limbs.

ELIGIBILITY:
Inclusion Criteria:

* Students will be screened for eligibility by testing their ability to perform a squat.

Exclusion Criteria:

* a recent (within one month) ankle sprain
* evidence of ankle instability
* cardiac condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in self-selected walking speed | Day 1 and 6 weeks
  Subjects will pick the speed they want to walk on the treadmill but will be blinded to their choice. The actual speed chosen will be recorded.

SECONDARY OUTCOMES:
Change in side-to-side difference in stance phase | Day 1 and 6 weeks
  Measurement of the change in the difference in single stance phase between the left foot and right foot.
Change in difference in step length from side-to-side | Day 1 and 6 weeks
  Measurement of the change in the difference in step length between the left foot and right foot

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Perle, DC, MS, Principal Investigator — University of Bridgeport
Locations (1):
- University of Bridgeport College of Chiropractic Human Performance Laboratory, Bridgeport, Connecticut, United States